CLINICAL TRIAL: NCT07320287
Title: A Randomized, Blinded, Controlled Trial to Evaluate Effects of Multi-strain Bacillus Spore Probiotic Supplements (LiveSpo PREG-MOM and LiveSpo CONSY) on Growth Metrics, Prevention of Functional Gastrointestinal Disorders, and Modulation of the Gut Microbiota in Cesarean-Delivered Neonates
Brief Title: Effects of Multi-strain Bacillus Spore Probiotics on Growth, Digestive Function, and Gut Microbiota in Cesarean-Delivered Neonates
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Collaborators: Hanoi Obstetrics and Gynecology Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TNLS.2025.NB
Record Dates: First submitted 2025-12-14; First posted 2026-01-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Functional Gastrointestinal Disorders (FGIDs); Weight Loss
Keywords: Cesarean-born Infants; Gut Dysbiosis; Bacillus spore
MeSH Terms: conditions — Gastrointestinal Diseases; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): The Placebo group receives reverse osmosis (RO) water with a dosage of 1 ampoule per day for 90 days.
  Interventions: Other: RO water
- Pregmom group (Experimental): The Pregmom group receives RO water plus B. subtilis, B. clausii, and B. coagulans at 3 billion CFU/5 mL (LiveSpo PREG-MOM) with a dosage of 1 ampoule per day for 90 days.
  Interventions: Combination Product: LiveSpo PREG-MOM
- Consy group (Experimental): The Consy group receives RO water plus B. subtilis, B. clausii, and B. coagulans at 4 billion CFU/5 mL (LiveSpo CONSY) with a dosage of 1 ampoule per day for 90 days.
  Interventions: Combination Product: LiveSpo CONSY

INTERVENTIONS:
Other: RO water — RO water (Aquafina, PepsiCo) produced under ISO 9001:2015 and ISO 22000:2018 standards. The RO water ampoules are produced using a similar process as the LIVESPO PREG-MOM/CONSY but contain 5 mL of high-quality RO water from Aquafina.
  Arms: Placebo group
Combination Product: LiveSpo PREG-MOM — LiveSpo PREG-MOM has a registration number 7695/2020/ĐKSP issued by the Food Safety Department of the Ministry of Health in Vietnam.
  Arms: Pregmom group
Combination Product: LiveSpo CONSY — LiveSpo CONSY has a registration number 4165/2020/ĐKSP issued by the Food Safety Department of the Ministry of Health in Vietnam.
  Arms: Consy group

SUMMARY:
Infants born by cesarean section commonly show early weight loss and slower recovery of birth weight, together with characteristic patterns of gut microbiota dysbiosis marked by reduced Bifidobacterium and Bacteroides and increased Proteobacteria. This early microbial alteration has been associated with functional gastrointestinal disorders (FGIDs), including colic, regurgitation, and changes in stool frequency and consistency, which may in turn affect early growth and overall gastrointestinal functioning. Probiotic supplementation is considered a safe and feasible strategy to support microbial restoration and improve digestive function during the first months of life.

In this study, researchers propose that daily supplementation with multi-strain Bacillus spore probiotics may help support healthy early growth, reduce functional gastrointestinal symptoms, and promote a more balanced gut microbiota in cesarean-delivered infants.

The objective of this study is to evaluate the safety and efficacy of two oral probiotic formulations, LiveSpo PREG-MOM and LiveSpo CONSY, containing multi-strain B. subtilis ANA46, B. clausii ANA39, and B. coagulans ANA40 at respective 3 and 4 billion colony-forming units (CFU)/5 mL ampoule, administered 1 ampoule daily, during the first 90 days of life. The study examines effects on growth, digestive symptoms, immune markers, and microbial composition.

Study Design: This randomized, blind, controlled clinical trial will enroll 180 healthy full-term cesarean-born infants at Hanoi Obstetrics and Gynecology Hospital.

Intervention Description: Participants will be randomly assigned to three groups (n = 60 each). All groups will receive one 5-mL ampoule daily for 90 days: LiveSpo PREG-MOM, LiveSpo CONSY, or placebo. Stool samples will be collected at several follow-up time points to assess digestive health and microbial development. All products will be provided in blinded and coded packaging to maintain objectivity.

Study Duration: 12 months

DETAILED DESCRIPTION:
Infants delivered by cesarean section commonly experience early differences in feeding and distinct patterns of gut microbial development compared with infants born vaginally. Because cesarean delivery limits contact with maternal vaginal microbiota, which is an important source of early microbial transfer, these infants often show delayed establishment of key early colonizers. Multiple cohort studies have documented lower abundances of beneficial genera such as Bifidobacterium and Bacteroides, along with relatively higher proportions of Proteobacteria during the first months of life. This shift in microbial composition has been associated with functional gastrointestinal symptoms in early infancy, including regurgitation, colic, abdominal discomfort, and changes in stool frequency and consistency. Such symptoms can affect feeding patterns, contribute to variations in weight gain, and influence overall gastrointestinal functioning during the neonatal period. As cesarean delivery rates continue to rise in Vietnam, there is increasing interest in supportive approaches that may help promote gastrointestinal functioning and healthier gut microbial development in this group.

Probiotic supplementation during early infancy has been explored as a potential strategy to support gut microbial maturation. Spore-forming Bacillus strains, belonging to safe B. subtilis, B. clausii, and B. coagulans species, are notable for their stability and ability to survive passage through the digestive tract. These characteristics allow them to reach the intestine in viable form, where they may interact with the developing gut ecosystem. Prior pediatric studies of Bacillus preparations have reported favorable safety profiles and signals of benefit for digestive conditions, although findings vary depending on strain and study design. Multi-strain products may offer complementary biological functions, providing broader support for the developing gut environment.

Based on this scientific background, the present study has been designed to evaluate two oral Bacillus spore probiotic formulations of B. subtilis ANA46, B. clausii ANA39, and B. coagulans ANA40, LiveSpo PREG-MOM (3 billion spores per 5 mL) and LiveSpo CONSY (4 billion spores per 5 mL), in cesarean-delivered infants. The study aims to evaluate whether daily supplementation during the first 90 days of life influences early growth trajectories, the occurrence of functional gastrointestinal disturbances, immune indicators in stool, and the development of gut microbial communities. The study will also assess the presence of probiotic spores in stool as an indicator of product use compliance.

This investigation is a randomized, blind, controlled clinical trial conducted at Hanoi Obstetrics and Gynecology Hospital. A total of 180 healthy full-term infants (38-40 weeks' gestation) delivered by cesarean section will be enrolled after parental consent. Eligible infants will be randomly assigned in equal numbers to one of three groups: Placebo (RO water), Pregmom (LiveSpo PREG-MOM), or Consy (LiveSpo CONSY). Randomization will use permuted blocks to help maintain balanced allocation across groups, and all products will be provided in identical coded ampoules to ensure blinding of families, clinical staff, and laboratory personnel.

Participants will receive one 5-mL ampoule of the assigned product once daily for 90 days. Clinical assessments will be performed at baseline and on days 2, 9, 30, 60, and 90. These assessments include measurements of weight, length, and head circumference, along with documentation of digestive patterns such as stool frequency, stool characteristics, regurgitation…, using structured observation tools suitable for young infants.

Stool samples will be collected at days 0, 2, 9, 30, 60, and 90 for laboratory evaluation. Real-time polymerase chain reaction (PCR) assays will be used to detect spores of B. subtilis, B. clausii, and B. coagulans, providing information on product exposure in the probiotic groups and verifying the absence of these strains in the placebo group. Stool samples collected on days 0, 9, and 30 will undergo enzyme-linked immunosorbent assay (ELISA)-based measurement of immune-related indicators, including pro- and anti-inflammatory cytokines, calprotectin, and immunoglobulin A (IgA), which may reflect aspects of intestinal immune activity. To investigate early microbial development, a subset of approximately 10-15 infants per group will undergo 16S ribosomal ribonucleic acid (rRNA) gene sequencing on stool samples collected at day 0 and day 30.

All data will be recorded in study-specific case report forms or electronic case report forms. Statistical analyses appropriate for categorical and continuous variables, as well as repeated measurements, will be applied according to the overall study objectives. The intervention period, scheduled follow-up visits, and data analysis will be completed within the 12-month study timeline.

Through the combined evaluation of growth patterns, digestive observations, immune indicators in stool, and microbiota profiles, this study aims to provide comprehensive evidence on the potential role of multi-strain Bacillus spore probiotics as a supportive option for infants born by cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term neonates delivered by cesarean section.
* Infants were born at term, ranging from 38 to 40 weeks' gestation.
* Birth weight appropriate for gestational age (AGA), defined as between the 10th and 90th percentiles for gestational age (≥P10 and ≤P90).
* The infant's parent(s) or legal guardian(s) provide written informed consent and agree to comply with study procedures.

Exclusion Criteria:

For the neonate:

* Multiple births (twins, triplets, etc.)
* Birth weight outside the appropriate-for-gestational-age range: small for gestational age (SGA, < P10) or large for gestational age (LGA, > P90).
* Major congenital abnormalities affecting the hematologic, hepatobiliary, cardiovascular, renal/urinary, or gastrointestinal systems; severe inborn errors of metabolism; or suspected primary immunodeficiency.
* Prior exposure to systemic or enteral antibiotics (oral, IV, or IM) before the baseline assessment.
* Known allergy or intolerance to any component of the investigational product.
* Concurrent participation in another interventional clinical trial.
* The investigators judge the neonate to be unsuitable for participation.
* Parent(s) or legal guardian(s) who do not comply with study requirements or refuse to sign the informed consent.

For the mother:

* Mother diagnosed with a serious or unstable medical condition involving the hepatobiliary, renal/urinary, cardiovascular, respiratory, endocrine/metabolic, or psychiatric systems.
* Mother who intends to use, or is prescribed, any other probiotic/prebiotic product for herself or the infant during the study period.

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-09-07 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Change in stool frequency | Days 0, 2, 9, 30, 60, and 90
  Change in daily stool frequency compared with baseline (day 0). Measurements at days 2, 9, 30, 60, and 90; days 2 and 9 serve as early supplementary timepoints.
Change in stool consistency (Diapered Infant Stool Scale score) | Days 0, 2, 9, 30, 60, and 90
  Change in stool consistency using the Diapered Infant Stool Scale (type 1-type 5) compared with baseline (day 0). Measurements at days 2, 9, 30, 60, and 90; days 2 and 9 serve as early supplementary timepoints.
Change in regurgitation | Days 0, 2, 9, 30, 60, and 90
  Change in regurgitation assessed by both frequency (number of regurgitation episodes per day) and severity (caregiver-reported severity), compared with baseline (day 0). Measurements will be obtained at days 2, 9, 30, 60, and 90; days 2 and 9 serve as early supplementary timepoints.
Change in crying episodes | Days 0, 2, 9, 30, 60, and 90
  Change in the number of crying episodes per day compared with baseline (day 0). Measurements at days 2, 9, 30, 60, and 90; days 2 and 9 serve as early supplementary timepoints.

SECONDARY OUTCOMES:
Change in infant body weight | Days 0, 2, 9, 30, 60, and 90
  Change in infant body weight (kg), and expressed as age-appropriate Z-scores based on WHO growth standards. Measurements at days 2, 9, 30, 60, and 90 will be compared with baseline (day 0).
Change in infant body length | Days 0, 30, 60, and 90
  Change in infant body length (cm), and expressed as age-appropriate Z-scores based on WHO growth standards. Measurements at days 30, 60, and 90 will be compared with baseline (day 0).
Change in infant head circumference | Days 0, 30, 60, and 90
  Change in infant head circumference (cm) and expressed as age-appropriate Z-scores based on WHO growth standards. Measurements at days 30, 60, and 90 will be compared with baseline (day 0).
Immune indicators in stool (cytokines and IgA) | Days 0, 9, and 30
  Changes in immune indicators measured in stool samples, including concentrations of selected pro-inflammatory and anti-inflammatory cytokines (for example, IL-1β, TNF-α, IL-6, IL-8, IL-10, IL-17) (µg/mL) and secretory IgA (µg/mL). Values at days 9 and 30 will be compared with baseline (day 0)
Gut microbiota composition | Days 0 and 30
  Changes in gut microbiota composition assessed by 16S rRNA gene sequencing of stool infants samples. Outcomes include diversity indices and relative taxonomic composition at major taxonomic levels (for example, phylum, family, genus) at day 30 compared with day 0

OTHER OUTCOMES:
Fecal calprotectin levels | Days 0, 9, and 30
  Changes in fecal calprotectin concentrations as an exploratory marker of intestinal inflammation, with values at days 9 and 30 compared with baseline.
Use of antibiotics during the study period | Day 0 to Day 90
  Use of systemic antibiotics over the 90-day follow-up, including the proportion of infants receiving at least one antibiotic course or/and the number of antibiotic courses per infant or/and the duration (days) of each antibiotic course. Information is collected at scheduled follow-up visits and summarized across the entire study period.
Detection of probiotic Bacillus spores in stool | Day 0 to Day 90
  Presence of B. subtilis, B. clausii, and B. coagulans spores in stool as determined by real-time PCR, used as an exploratory indicator of exposure to the assigned probiotic products and adherence to the intervention across follow-up timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Hung T Mai, PhD, Principal Investigator — Hanoi Obstetrics and Gynecology Hospital; Chuong C Nguyen, Study Chair — Hanoi Obstetrics and Gynecology Hospital; Anh TV Nguyen, Assoc.Prof.PhD, Study Chair — Anabio R&D
Locations (1):
- Hanoi Obstetrics and Gynecology Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e., a material transfer agreement) are prerequisites to the sharing of data with the requesting party
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted 9 months after article publication and will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research. It will be provided following the review and approval of a study protocol, informed consent form (ICF), clinical study report (CSR), and Statistical Analysis Plan (SAP). For more information or to submit a request, please get in touch with anabio.rd2021@gmail.com

REFERENCES:
- [Background] Long G, Hu Y, Tao E, Chen B, Shu X, Zheng W, Jiang M. The Influence of Cesarean Section on the Composition and Development of Gut Microbiota During the First 3 Months of Life. Front Microbiol. 2021 Aug 18;12:691312. doi: 10.3389/fmicb.2021.691312. eCollection 2021. PMID 34489887
- [Background] Kelly NM, Keane JV, Gallimore RB, Bick D, Tribe RM. Neonatal weight loss and gain patterns in caesarean section born infants: integrative systematic review. Matern Child Nutr. 2020 Apr;16(2):e12914. doi: 10.1111/mcn.12914. Epub 2019 Nov 27. PMID 31777183
- [Background] Ianiro G, Rizzatti G, Plomer M, Lopetuso L, Scaldaferri F, Franceschi F, Cammarota G, Gasbarrini A. Bacillus clausii for the Treatment of Acute Diarrhea in Children: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Nutrients. 2018 Aug 12;10(8):1074. doi: 10.3390/nu10081074. PMID 30103531
- [Background] Gong Y, Zhong H, Wang J, Wang X, Huang L, Zou Y, Qin H, Yang R. Effect of Probiotic Supplementation on the Gut Microbiota Composition of Infants Delivered by Cesarean Section: An Exploratory, Randomized, Open-label, Parallel-controlled Trial. Curr Microbiol. 2023 Sep 15;80(11):341. doi: 10.1007/s00284-023-03444-4. PMID 37712964
- [Background] Delfino E, Peano L, Wetzl RG, Gianni ML, Netto R, Consales A, Bettinelli ME, Morniroli D, Vielmi F, Mosca F, Montagnani L. Newborn Weight Loss as a Predictor of Persistence of Exclusive Breastfeeding up to 6 Months. Front Pediatr. 2022 Apr 7;10:871595. doi: 10.3389/fped.2022.871595. eCollection 2022. PMID 35463877
- [Background] Colom J, Freitas D, Simon A, Brodkorb A, Buckley M, Deaton J, Winger AM. Presence and Germination of the Probiotic Bacillus subtilis DE111(R) in the Human Small Intestinal Tract: A Randomized, Crossover, Double-Blind, and Placebo-Controlled Study. Front Microbiol. 2021 Aug 2;12:715863. doi: 10.3389/fmicb.2021.715863. eCollection 2021. PMID 34408741
- [Background] Bernardeau M, Lehtinen MJ, Forssten SD, Nurminen P. Importance of the gastrointestinal life cycle of Bacillus for probiotic functionality. J Food Sci Technol. 2017 Jul;54(8):2570-2584. doi: 10.1007/s13197-017-2688-3. Epub 2017 May 23. PMID 28740315